CLINICAL TRIAL: NCT07161063
Title: A Program Evaluation of the Brief Family Therapy Program in the York University Psychology Clinic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Principal Investigator, Heather Prime, Associate Profesor, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e2025-244
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Family Relationships; Child Mental Health; Coparenting
Keywords: Brief Family Therapy; Family Systems; Coparenting; Feasibility Study; Implementation Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Family Therapy Program (Experimental): Families will take part in a four-session video-feedback intervention.
  Interventions: Behavioral: Brief Family Therapy Program

INTERVENTIONS:
Behavioral: Brief Family Therapy Program — The Lausanne Family Play - Brief is a video-feedback intervention adapted for families seeking support for a child two to nine years old with a mental health challenge. Feedback focuses on engagement, teamwork, conflict, and child-focused issues.
  Other Names: LFP-B; Lausanne Trilogue Play-Brief (LTP-B)

SUMMARY:
Background. Children are vulnerable to mental health challenges during development. Given that youth are reliant on their parents for support, understanding the child's symptoms within the family context is critical for promoting positive change. This proposal focuses on "systemic therapy", or family-based therapy, which seeks to enhance children's mental health by improving the relationships and communication between family members (1). Most family-based therapies for treating child mental health problems are intense in duration and frequency (2), which is a barrier to access for many families. Shorter-term family therapies or what will be referred to hereafter as brief family-based therapies are effective in treating a variety of child symptoms, while also minimizing participant burden and therapy dropout (3). One type of brief family-based therapy model is the Lausanne Family Play - Brief (LFP-B), a three-session service that utilizes a play-based family observational assessment with video feedback to draw attention to and catalyze change in challenging family interactions. The LFP has been widely researched as a clinical assessment tool and has been implemented as a brief family-based therapy program (4). The current project represents the implementation and evaluation of the program in the York University Psychology Clinic (YUPC), which services children, adults, couples, and families in the Greater Toronto Area (and Ontario, broadly). The current study will be the first to evaluate the implementation, acceptability, and effectiveness of the LFP-B as a clinic service. Objectives. The aim of this project is to evaluate the LFP-B as a brief family-based clinical service offered in the YUPC. The first objective is to explore program acceptability for both clients and therapists. The investigators are interested in whether clients and therapists are satisfied with this clinical service and its processes. The second objective is to assess program effectiveness, specifically whether coparenting, family functioning, and child mental health problems improve across the course of the program and in the months following. Importance. Brief therapies with a systemic lens can increase cost-effectiveness, accessibility, and treatment retention. They also have potential to fill an apparent gap in service needs as up to three-quarters of youth with psychological concerns never receive treatment (5). Thus, brief services can provide more timely access to mental health care in Canada which have potential for reducing wait times, preventing further deterioration in mental health, and avoiding more intensive and expensive higher levels of care (e.g., acute inpatient mental health services; (6)). The LFP-B has potential to be widely used as a brief family-based therapy program with Canadian families to support child and family functioning in a timely and non-intensive manner.

ELIGIBILITY:
Inclusion Criteria:

* Both primary caregivers are over age 18 years
* Families living in Ontario, Canada
* Primary caregivers endorses caring for a child between 2 to 9 years old with a mental health challenge (e.g., anxiety, low mood, behavioural challenges) or mild/moderate levels of family distress
* Both caregivers and child agree to participate
* Family must have access to a screen (phone, tablet, computer) and internet for virtual services and recording.

Exclusion Criteria:

- Families seeking care for child who is at imminent risk of harm to self or others

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Referral Sources | Week 0
  Where participants heard about the program (e.g., social media, YUPC, employee, friend)
Participants Enrolled Per month | Week 0
  Number of participants enrolled per month
Service Enrollment Rate | Week 0
  Proportion of participants offered the service versus those who actually sign up
Reasons for Non-Enrollment | Week 0
  Reasons for not joining the service for those who were offered it (e.g., scheduling multiple caregivers, desire for child-focused treatment, cost, time commitment, etc.)
Waitlist Duration | Week 0
  Time in days from initial intake call to first phone call with clinician
Participant Education | Week 1
  The percentage of participants with less than or equal to a high school degree.
Geographic Reach | Week 0
  Cities/towns in Ontario families accessing the program reside
Retention | Week 8
  The percentage of participants who remain in study until the end of the follow up session.
Service Uptake | Week 8
  The percentage of participants reporting some reflection about coparenting outside of sessions.
Client Acceptability | Week 8
  Looking for the percentage of participants reporting at least 'good' on 80 % or more indicators on an Implementation Acceptability Scale that will assess attitude, burden, perceived effectiveness, and ethicality. Minimum score=7, maximum score=35. Higher scores correspond to better outcomes.
Clinician Acceptability | Week 8
  Looking for the percentage of clinicians reporting at least 'good' on 80 % or more indicators on an Implementation Acceptability Scale that will assess attitude, burden, perceived effectiveness, and ethicality. Minimum score=7, maximum score=35. Higher scores correspond to better outcomes.
Working Alliance Inventory | Longitudinal change across week 1 to week 8
  Exploratory for pattern of scores across the intervention on a Working Alliance Inventory Scale that will assess client perceptions of goals, tasks, and bonds during intervention. Scores range from 12-60 with higher scores representing greater self-reported alliance.
Pre-Post Change in Parent Reported Coparenting Relationship | Pre-post change from week 1 to week 8
  Using the Coparenting Scale-Revised (McHale, 1999; unpublished manuscript). Minimum score=18, maximum score=90. Higher scores correspond to a greater frequency of outcomes.

SECONDARY OUTCOMES:
Pre-Post Change in Parenting Stress | Pre-post change from week 1 to week 8
  Using the Parental Stress Scale (PSS; Berry & Jones, 1995). Minimum score=18, maximum score=90. Higher scores correspond to worse outcomes (i.e., more stress).
Pre-Post Change in Child Reported Coparenting Relationship | Pre-post change from week 2 to week 8
  Using the Child Perspectives on the Coparenting Relationship - Revised (created based on McHale's 1999 Coparenting Scale - Revised). Minimum score=7, maximum score=21. Higher scores correspond to a greater frequency of outcomes.
Pre-Post Change in Parent and Child Family Adjustment | Pre-post change from week 1 to week 8
  Using the Parenting and Family Adjustment Scale (PAFAS; Sanders & Morawska, 2010). Minimum score=0, maximum score=90. Higher scores correspond to worse outcomes (i.e., higher levels of dysfunction).
Pre-Post Change in Child Emotional Distress (i.e., Anger, Anxiety, and Depressive Symptoms) | Pre-post change from week 0 to week 8
  Using the subscales of the Emotion Distress scale of the Patient-Reported Outcomes Measurement Information System (NIH) Parent Proxy Domains (ages 5-17) or Early Childhood Parent Report (ages 1-5). Ages 5-17 minimum score = 19, maximum score = 120 Ages 1-5 minimum score = 24, maximum score = 120. Higher scores correspond to worse outcomes (i.e., more emotional distress).
Pre-Post Change in Child Externalizing Problems | Pre-post change from week 1 to week 8
  Using the Externalizing Problems subscale of the Behavior and Feelings Survey (BFS) Caregiver Report Form (Weisz et al., 2019). Minimum score=0, maximum score=24. Higher scores correspond to worse outcomes (i.e., more behavioural problems).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Prime, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schleider JL, Weisz JR. Little Treatments, Promising Effects? Meta-Analysis of Single-Session Interventions for Youth Psychiatric Problems. J Am Acad Child Adolesc Psychiatry. 2017 Feb;56(2):107-115. doi: 10.1016/j.jaac.2016.11.007. Epub 2016 Nov 25. PMID 28117056
- [Background] Graziano PA, Ros-Demarize R, Hare MM. Condensing parent training: A randomized trial comparing the efficacy of a briefer, more intensive version of Parent-Child Interaction Therapy (I-PCIT). J Consult Clin Psychol. 2020 Jul;88(7):669-679. doi: 10.1037/ccp0000504. Epub 2020 Apr 30. PMID 32352803
- [Background] Philipp DA, Prime H, Darwiche J. An ultra-brief systemic intervention to address child mental health symptomatology. Fam Process. 2023 Jun;62(2):469-482. doi: 10.1111/famp.12875. Epub 2023 Mar 23. PMID 36959726
- [Background] Carr, A. (2019). Family therapy and systemic interventions for child-focused problems: the current evidence base. Journal of Family Therapy, 41(2), 153-213. https://doi.org/10.1111/1467-6427.12226
- [Background] Karam, E. A., Blow, A. J., Wampler, K. S., Seedall, R. B., & Miller, R. B. (2020). Common Factors Underlying Systemic Family Therapy. In The Handbook of Systemic Family Therapy (pp. 147-169). John Wiley & Sons, Ltd. https://doi.org/10.1002/9781119438519.ch7